CLINICAL TRIAL: NCT03619278
Title: A Phase I/IIa, Randomised Study to Evaluate the Safety and the Effectiveness of a Combination of Therapeutic Vaccine, Broadly Neutralising Antibody (10-1074), and the Latency Reversing Agent Romidepsin to Achieve a Remission of HIV Infection in Chronically HIV-infected Participants Under Stable Combined Antiretroviral Therapy.
Brief Title: Evaluating a Combination of Immune-based Therapies to Achieve a Remission of HIV Infection
Acronym: HIVACAR
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The clinical trial was discontinued prior to initiation due to the withdrawal of the vaccine manufacturer (etherRNA) from the research consortium. As a result, the study could not proceed as originally planned.
Sponsor: Judit Pich (Other)
Responsible Party: Sponsor-Investigator, Judit Pich, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-000566-30
Record Dates: First submitted 2018-03-14; First posted 2018-08-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIVACAR (Experimental): Participants will receive 5 vaccines of personalized RNA vaccine (HIVACAR01), 2 dose of 10-1074 antibodies and 3 doses of romidepsin
  Interventions: Other: HIVACAR
- Placebo (Placebo Comparator): Participants will receive 5 doses of placebo, 2 doses of 10-1074 antibodies and 3 doses of romidepsin
  Interventions: Other: placebo

INTERVENTIONS:
Other: HIVACAR — Participants will receive 5 vaccines of personalized RNA vaccine (HIVACAR01), 2 doses of 10-1074 antibodies and 3 doses of romidepsin
  Arms: HIVACAR
Other: placebo — Participants will receive 5 vaccines of placebo of HIVACAR01, 2 doses of 10-1074 antibodies and 3 doses of romidepsin
  Arms: Placebo

SUMMARY:
A phase I/IIa, multinational, multicentric (IDIBAPS, IRSICAIXA, AARHUS, VUB, APHP), randomised, balanced by centre (to include participants from the 4 arms), open-label, controlled clinical trial. Each participant will be followed up a different time according to study arm: a minimum of 38 weeks in arm I, 31 weeks in arm II, 54 weeks in arm III and 26 weeks in the arm 4. The study duration will be 104 weeks from inclusion of the first participant.

Participants will be randomised to one of the following 4 arms:

* Arm 1 (study): 14 participants will receive 3 vaccines of HIVARNA01.3 prime, 2 MVA-vectored vaccine boosts, 1 dose of 10-1074 antibodies and 3 doses of romidepsin
* Arm 2 (study): 14 participants will receive 5 vaccines of HIVARNA01.3, 1 dose of 10-1074 antibodies and 3 doses of romidepsin
* Arm 3 (study): 14 participants will receive 5 vaccines of personalized RNA vaccine (HIVACAR01), 1 dose of 10-1074 antibodies and 3 doses of romidepsin
* Arm 4 (control): 14 participants 1 dose of 10-1074 antibodies and 3 doses of romidepsin

ELIGIBILITY:
Inclusion Criteria:

1. Between ≥ 18 to <60 years of age
2. Voluntarily signed informed consent
3. Male, or female with negative pregnancy test prior to enrolment
4. Proven HIV-1 infection (with positive antibodies against HIV-1 and a detectable plasma HIV-1 RNA before cART)
5. Must be on stable treatment with cART for at least 18 months (cART is defined as an antiretroviral regimen consisting of at least three registered antiretroviral agents; periods of mono/dual antiretroviral therapy if not first time therapy and confirmed viral suppression during these periods of mono/dual therapy are permitted)
6. Nadir CD4+ cell counts must be above or equal to 350 cells/µl, 2-3 occasional determinations below 350 cells/μl are allowed.
7. Current CD4+ cell count must be at least 450 cells/µl
8. HIV-RNA must be below 50 copies/ mL for the last 12 months prior to inclusion, during at least two measurements (occasional so called 'blips' up to 500 copies/mL are permitted)
9. If male or female of childbearing potential willing to take correct contraceptive measures:

   1. If heterosexually active female; using an effective method of contraception from 14 days prior to the first vaccination until at least 12 weeks after the last vaccination; all female volunteers must be willing to undergo urine or serum pregnancy tests at time points specified in the Schedule of Procedures.
   2. If heterosexually active male; willing to use an effective method of contraception or agree on the use of an effective method of contraception by his partner from the day of the first vaccination until 12 weeks after the last vaccination.
10. If sexually active, willing to use a reliable method of reducing the risk of transmission to their sexual partners during treatment interruption (which could include pre-exposure prophylaxis [PrEP] for their sexual partners)

Exclusion Criteria:

1. Treatment with a non-cART regimen of antiretroviral agents prior to the start of any antiretroviral regimen
2. History of a CDC class C event (see Appendix IV)
3. Women of childbearing potential with a positive pregnancy test, or participants (male or female) who wish to plan a pregnancy during the trial period.
4. Active opportunistic infection, or any active infection or malignancy within 30 days prior to screening visit
5. Therapy with immunomodulatory agents, including cytokines (e.g. IL2) and gamma globulin, or cytostatic chemotherapy within 90 days prior to screening visit
6. Use of anti-coagulant medication
7. Use of any investigational drug during the 90 days prior to study entry
8. Previous antiretroviral therapy failure and/or mutations conferring genotypic resistance to antiretroviral therapy
9. Participants with severe cardiovascular diseases or long QT interval
10. Active hepatitis C virus
11. Hepatitis B infection
12. Treatment with strong inhibitors or inducers of CYP3A4, except protease inhibitors for HIV treatment (see protocol section 5.7); if in treatment of protease inhibitors for HIV not willing to change inhibitor protease for an integrase inhibitor during the study.
13. Any known allergy or intolerance to any of the study drugs or excipient
14. Protein egg allergy
15. Known past history of clinical Epstein-Barr Virus (EBV) infection or recurrent herpes zoster
16. Hematologic abnormalities ≥Grade 1
17. Potassium or magnesium levels outside the upper limit of normal (ULN) and lower limit of normal (LLN)
18. History of autoimmune disorders as multiple sclerosis.
19. Any other condition which, in the opinion of the investigator, may interfere with the evaluation of the study objectives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or above severe local , systemic, clinical or laboratory adverse event t | 12 days (28 days after each inmuisation)
  Local adverse events may be pain, cutaneous reactions including induration and systemic emperature, chills, headache, nausea, vomiting, malaise, and myalgia. Clinical and laboratory must be confirmed at examination or on repeat testing respectively. Any adverse event attributable to the combination therapy leading to discontinuation of the study treatmen

SECONDARY OUTCOMES:
Proportion of participants who maintain an undetectable viral load | 12 weeks (after discontinuation of antiretroviral therapy)
  defined as a viral load below the threshold of 50 copies/ml
Percentage of participants with control of viral load below detectable level | 24 weeks (after discontinuation of antiretroviral therapy)
Change from baseline in total proviral HIV-1 DNA per 10^6 CD4+ T cells. | up to 51 weeks
Change from baseline in integrated proviral HIV-1 DNA per 10^6 CD4+ T cells. | up to 51 weeks
Change from baseline in HIV-1 transcription. | up to 39 weeks
  According to CA US HIV-1 RNA measured in unfractionated CD4+ T cells
Change in plasma HIV-1 RNA from baseline | up to 39 weeks
Breadth and magnitude of CD4+ HIV-specific T cell responses measured by IFN-gamma ELISPOT compared with baseline. | up to 27 weeks
Breadth and magnitude of CD8+ HIV-specific T cell responses measured by IFN-gamma ELISPOT compared with baseline. | up to 27 weeks
Breadth and magnitude of CD4+ HIV-specific T cell responses measured by Intra-cellular cytokine staining-ICS in the study arms as compared with baseline. | up to 27 weeks
Breadth and magnitude of CD8+ HIV-specific T cell responses measured by Intra-cellular cytokine staining-ICS in the study arms as compared with baseline. | up to 27 weeks
Change from baseline in CD8+ T-cell HIV suppressive capacity. | up to 51 weeks
Change from baseline in T cell activation markers | up to 29 weeks
Change from baseline in T cell activation markers | 3 weeeks
Change from baseline in T cell activation markers | up to 24 weeks
Change from baseline in T cell subset distribution | up to 29 weeks
Change from baseline in T cell subset distribution | 14 weeks
Change from baseline in T cell subset distribution | up to 27 weeks
Change from baseline in PD-1 expression | up to 51 weeks
Evaluate fecal microbiome | baseline and at week 14
Characterise viral escape from vaccine-induced immune T cell responses | up to 51 weeks
  Comparison of viral sequences pre-cART and rebounding after cART interruption
Analysis of changes in sensitivity to neutralisation by 10-1074 of rebounding viruses after cART interruption to identify neutralisation escape mutants. | up to 51 weeks
To evaluate mRNA expression profiles in whole PBMC at baseline | at first romidepsin administration and 14 and 26 weeks after first romidepsin administration

IPD SHARING:
Plan to Share IPD: Undecided